CLINICAL TRIAL: NCT03029741
Title: A Phase I Study To Assess The Absolute Bioavailability Of A Single Oral Dose Of AZD0284 And To Assess The Pharmacokinetics Of A Single Intravenous Microdose Of [14C]AZD0284 In Healthy Subjects.
Brief Title: Bioavailability of AZD0284 and IV Microtracer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7800C00002; 2016-004260-19 (EudraCT Number)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Plaque Psoriasis Vulgaris
MeSH Terms: interventions — AZD-0284

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bioavailability of AZD0284 (Experimental): To assess the absolute bioavailability of a single oral dose of AZD0284 in healthy subjects.
  To assess the pharmacokinetics (PK) of a single intravenous (IV) microdose of [14C]AZD0284 in healthy subjects.
  Interventions: Drug: AZD0284; Drug: [14C]AZD0284

INTERVENTIONS:
Drug: AZD0284 — Subjects will receive a single oral dose of 4 to 120 mg AZD0284 oral suspension 5 mg/mL in the fasted state
Drug: [14C]AZD0284 — Following administration of the AZD0284 oral suspension subjects will receive an IV infusion of 20 μg [14C]AZD0284 solution

SUMMARY:
The Sponsor is developing the study drug, AZD0284, for the potential treatment of Plaque psoriasis. Psoriasis is a skin condition that causes red, flaky, crusty patches of skin covered with silvery scales. It occurs when skin cells are replaced more quickly than usual. The seriousness of psoriasis varies greatly from person to person. For some people it is a minor irritation, but for others it can have a major impact on their quality of life. .

The purpose of the study is to determine how much of AZD0284 is taken up by the body. The safety and tolerability of the drug will also be assessed. It is hoped that the study drug will improve the management of psoriasis.

DETAILED DESCRIPTION:
The study is a Phase I, single centre, open-label, non-randomized, single dose study performed in 6 healthy male subjects aged 18 to 65 years, inclusive. The study will assess the absolute bioavailability of a single oral dose of AZD0284 and the pharmacokinetics (PK) of a single intravenous (IV) microdose of [14C]AZD0284 in healthy male and female subjects. Oral AZD0284 and [14C] AZD0284 intravenous solution are referred to as the investigational products in this study.

A screening visit to assess the eligibility of the healthy male and female subjects will occur within 28 days of the administration of the investigational product. Screening assessments will include medical history, inclusion/exclusion criteria, demographic data, weight and height, vein assessment, physical examination, blood samples for haematology, clinical chemistry and virology, blood test to confirm post-menopausal status (if female and of non-childbearing potential), blood test to confirm no history of tuberculosis, urine sample for urinalysis, urine test for pregnancy (if female and of childbearing potential) drug screen, alcohol breath test, carbon monoxide (CO) breath test, heart monitoring using ECG, vital signs (blood pressure, heart rate) Study related procedures will only be performed after signing of the Informed Consent Form.

The healthy male and female subjects will be admitted to the study centre the day before administration of the investigational product (Day -1). On Day 1, subjects will be dosed with a single oral dose of 4 to 120 mg AZD0284 oral suspension (Regimen A) followed by 20 μg [14C]AZD0284 solution for IV infusion (Regimen B) beginning 3 hours after the oral dose has been administered. The IV microdose will be infused over 15 minutes and the end of the infusion is expected to be around the predicted tmax of Regimen A.

The subjects will remain in the study centre until the 48 hour post dose PK blood sample is obtained. A follow up visit will occur 5 to 7 days after dosing and will include PK and routine safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated, written informed
2. Healthy males or non-pregnant, non-lactating healthy females.
3. Age 18 to 65 years of age.
4. Suitable veins for cannulation or repeated venepuncture.
5. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria:

   * Post-menopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the postmenopausal range.
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
6. Body mass index of 18.0 to 30.0 kg/m2, inclusive, or, if outside the range, considered not clinically significant by the investigator, and weigh at least 50 kg and no more than 100 kg, inclusive.
7. Must be willing and able to communicate and participate in the whole study.
8. Must agree to use an adequate method of contraception

Exclusion

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results of the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
4. Subject who have increased risk of infection History and/or presence of tuberculosis (TB) positive result for IFN-y release assay (IGRA) (ie QuantiFERON TB-Gold). The test may be repeated if the initial test result is indeterminate.

   Is in a high-risk group for human immunodeficiency virus (HIV) infection within the last 6 months.

   Subjects with a disease history suggesting abnormal immune function in the judgement of the investigator. (This does not include mild allergy such as childhood asthma or eczema).
5. Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis, as judged by the investigator.
6. Any clinically significant abnormal findings in vital signs, as judged by the investigator.
7. Any clinically significant abnormal findings in 12-lead ECG, as judged by the investigator.
8. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or HIV results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Determination of absolute bioavailability of AZD0284 | PK blood samples: pre-dose, post oral dosing at hour, 0.5, 1, 2, 0, 0.5, 1, 2, 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5,3.75, 4, 5, 6, 7, 8, 9, 11, 12, 15, 24, 27, 36, 48 and 72.
  Absolute bioavailability of AZD0284 will be calculated from area under the plasma concentration versus time curve (AUC) of the oral dose of AZD0284 / AUC of the IV dose of [14C]AZD x IV dose/Oral dose x 100
Cmax for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0824 in terms of the maximum observed plasma concentration (Cmax) for [14C]AZD0284
Tmax for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the the time to maximum observed plasma concentration (Tmax) for [14C]AZD0284.
AUC(0-last) for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the area under the concentration-time curve from dosing to the last measurable concentration for [14C]AZD0284.
AUC(0-inf) for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms the area under the concentration-time curve from dosing extrapolated to infinity for [14C]AZD0284.
AUC%extrap for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the percentage of AUC(0-inf) extrapolated beyond the last measured for [14C]AZD0284.
lambda-z for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the terminal elimination rate constant calculated from the slope of the apparent elimination phase for [14C]AZD0284.
T1/2 for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the apparent terminal elimination half-life for [14C]AZD0284.
CL (total clearance) for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the terminal elimination rate constant calculated from the slope of the apparent elimination phase for [14C]AZD0284
Vz for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the volume of distribution at steady state for [14C]AZD0284.
Vss for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the volume of distribution at steady state for [14C]AZD0284.
MRT (mean residence time) for [14C]AZD0284 | PK blood samples:pre-dose, time relative to oral dosing at hour: 2.83, 2.92, 2.92, 3, 3.08, 3.17, 3.33, 3.5, 3.75, 4, 5, 6, 7, 8, 9, 11, 15, 27, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the IV dose of AZD0284 in terms of the mean residence time for [14C]AZD0284.
Cmax for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0824 in terms of the maximum observed plasma concentration (Cmax) for AZD0284.
Tmax for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the the time to maximum observed plasma concentration (Tmax) for AZD0284.
Tlag for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the elapsed time from dosing at which the analyte was first quantifiable in a concentration vs time profile for AZD0284.
AUC (0-last) for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the area under the concentration-time curve from dosing to the last measurable concentration for AZD0284.
AUC(0-inf) for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms the area under the concentration-time curve from dosing extrapolated to infinity for AZD0284.
AUC%extrap for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the percentage of AUC(0-inf) extrapolated beyond the last measured time point for AZD0284.
lambda-z for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the terminal elimination rate constant calculated from the slope of the apparent elimination phase for AZD0284.
T1/2 for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the apparent terminal elimination half-life for AZD0284.
CL/F for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the apparent total clearance for AZD0284.
Vz/F for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 , 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms of the apparent volume of distribution for AZD0284.
MRT for AZD0284 | PK blood samples: pre-dose, time relative to oral dosing at hour, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72.
  Pharmacokinetic (PK) profile of the oral dose of AZD0284 in terms the mean residence time for AZD0284.

SECONDARY OUTCOMES:
To collect further information about the safety and tolerability of AZD0284 by assessing physical examinations. | Targeted physical examination:screening, pre-dose, time relative to oral dosing at hour 72.
  Physical examination will be carried out by a fully registered physician at the clinical unit.
To collect further information about the safety and tolerability of AZD0284 by assessing telemetry | Continuous ECG monitoring will commence approximately 10 minutes before dosing commences until 24 hours after the oral dose.
  ECGs will be taken in the clinic by a trained research nurse or a trained clinical technician and reviewed by a physician.
To collect further information about the safety and tolerability of AZD0284 by assessing safety laboratory tests | Haematology and clinical chemistry:screening, pre-dose, time relative to oral dosing at hour 24 and 72, virology at screening.
  Collected by a research nurse or trained clinical technician at the clinical unit.
To collect further information about the safety and tolerability of AZD0284 by assessing vital signs | Blood pressure and pulse rate: screening, pre-dose, post oral dosing at hour 1, 2, 3, 4, 6, 8, 12, 24 and 72.
  Vital signs will be measured using manual and automated devices by trained staff at the clinical unit.
To collect further information about the safety and tolerability of AZD0284 by assessing 12 Lead Electrocardiogram (ECG) | ECGs: screening, pre-dose, post oral dosing at hour, 1, 2, 3, 4, 6, 8, 12, 24 and follow up.
  ECGs will be taken in the clinic by a trained research nurse or a trained clinical technician and reviewed by a physician.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, MRCS, Principal Investigator — Quotient Clinical Ltd, United Kingdom
Locations (1):
- Research Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No